CLINICAL TRIAL: NCT02191514
Title: Prehospital Management of Stroke Patients by Emergency Medical Services - an Evaluation of Emergency Medical Dispatch and Ambulance Personnel.
Brief Title: Prehospital Management of Stroke Patients by Emergency Medical Services
Status: Completed | Type: Observational
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: University of Copenhagen (Other); Bispebjerg Hospital (Other); Glostrup University Hospital, Copenhagen (Other); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Other Study IDs: EMS-2014-SV-01
Record Dates: First submitted 2014-06-30; First posted 2014-07-16 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Stroke
Keywords: Prehospital; EMS; EMD; Stroke; Dispatch
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Annually 12.000 people i Denmark suffer from a stroke. Treatment for ischemic stroke is available, but only 12% of stroke patients receive it.

The treatment is only available within a time frame of 4,5 hours from symptom onset, thus the Emergency Medical Services (EMS) is essential to fast and effective stroke treatment.

The aim of this study is:

1. To establish the rate of recognition of stroke symptoms by healthcare personnel in the EMD, ultimately aiming at optimizing performance, and identifying barriers for a fast and correct EMS-response.
2. To assess prehospital time consumption by ambulance personnel on the scene of a stroke, create a baseline for future comparison and generate explorative hypotheses for forthcoming interventions.

The overall aim of this study is, to ensure the best possible prehospital care for all stroke patients. The study will determine, if the EMD is at a high and international level in regards to stroke recognition, and if there is a potential to decrease on-scene time. This will serve as future comparison and have an effect on the structure and future education in the prehospital services, and potentially improve the outcome after acute ischemic stroke.

DETAILED DESCRIPTION:
Background:

Approximately 12.000 strokes occur in Denmark annually. The only evidence based pharmacological treatment of ischemic stroke is thrombolysis within a time-window of 4.5 hours from symptom onset(1). In 2012, 12% of patients with ischemic stroke in Denmark received thrombolysis treatment. The probability of a favourable 3-month outcome after stroke decreases with time from symptom onset to thrombolysis: the onset to needle time(2). Therefore, it is of the highest importance to identify potential targets for prehospital time reduction, and thereby reduce delay to definitive care.

Prompt recognition of stroke symptoms by both the EMD and ambulance personnel is a crucial step, as it provides access to fast track acute stroke services. In this context, the role of the EMS is essential, as contact to the hospital through EMS opposed to private transport is correlated to decreased onset-to-door time (3). EMS prenotification of the stroke centre is correlated to shorter door-to-evaluation time, door-to-needle time and onset-to-needle time(4). In Denmark EMS prenotification in acute stroke is well established.

According to Danish guidelines for treatment of acute stroke and transient ischaemic attack (TIA), prehospital diagnosis of stroke is improved by use of validated tests. No such is yet implemented in the Capital Region of Denmark.

Preliminary data shows that the mean time from the ambulance personnel arrives at the scene to they start the transport to the hospital ("on scene time") is 18 minutes in the Capital Region of Denmark. American guidelines suggest that on-scene-time should be less than 15 minutes in all cases (unless extenuating circumstances or extrication difficulties are present)(1), however the organisation of stroke care between Scandinavia and USA varies largely.

The aim of this study is:

1. To establish the rate of recognition of stroke symptoms by healthcare personnel in the EMD, ultimately aiming at optimizing performance, and identifying barriers for a fast and correct EMS-response.
2. To assess prehospital time consumption by ambulance personnel on the scene of a stroke, create a baseline for future comparison and generate explorative hypotheses for forthcoming interventions.

The study consists of 3 arms:

1. An epidemiological analysis of prospectively collected data from a 2-year period, in order to establish the rate of identification of stroke symptoms by healthcare personnel in the EMD.
2. A quantification and statistical analysis of on-scene-time in stroke patients, based on prospectively collected data from a registration form filled out by the ambulance personnel after responding to a stroke. The focus of the form is on time spent on predefined tasks aiming at assessing time consumption on the scene, and generating explorative hypotheses for forthcoming interventions.
3. Based on EMS data, the investigators will establish a baseline for on-scene-time and transportation time in patients admitted by fast track stroke service during a 6 months period, for future comparison and analyse data in conjunction with in-hospital delays.

Method for each arm:

1. The epidemiological analysis is based on prospectively collected data from the Danish Stroke Registry (DSR) and the National Patient Registry (NPR). In the DSR and NPR, ICD-10-codes are linked to the Danish personal identification number, a unique number for every Danish citizen. The investigators shall compare ICD-10 codes from DSR and NPR with dispatch codes from the EMS database, to determine the amount of diagnosed stroke patients recognized during the emergency call. The date of the incident report from the EMS will be matched with the admission date correlated to the discharge ICD-10 code, in case a patient has been admitted more than once.
2. To quantify and analyse prehospital time consumption, the investigators will develop a registration form for the ambulance personnel to fill out after responding to a stroke patient.

   This registration form will include registration of time intervals spent on:
   * Clinical tasks; including prior medical history, clinical examination and measurement of vital parameters
   * Communication in relation to prenotification of the stroke centre
   * Mobilization of the patient and on-scene conditions
   * Patient preparation; including IV-accesses and 12-lead ECG

   As well as information regarding:
   * Patient preparation; including IV-accesses and 12-lead ECG
   * Language/communication barriers
   * Specifications of the ambulance (operator, level of education)
   * Patient/relative related conditions
   * Visitation to acute stroke fast track

   Statistical analyses:

   Poisson regression analyses will be made with over dispersion taken into account, in order to identify specific time intervals and tasks correlated to extended or decreased total on-scene-time. This model yields distributions similar to previously collected data.

   A power calculation has been made, based on this distribution and the assumption that a clinically relevant difference, is defined as any time interval in cases considered as having a high on-scene-time, (>15 min.) being twice the amount than in cases considered as having a low on-scene-time (≤15 min.). This has shown an estimated demand of 500 registration forms in order to achieve a power of 0,8 with a 5% two-sided confidence interval.
3. The establishment of on-scene-times and transportation-times will be made by extracting specific time points (e.g. ambulance arrival at the scene, departure towards hospital and arrival at hospital) from the EMS database during a 6 months period, and analysed in conjunction with data on in-hospital delays.

The stroke centres will provide Danish personal identification numbers for patients referred to the stroke centres as well as door-to-needle times and treatment decisions in order to determine if there is a correlation be-tween recognition and treatment decisions in stroke fast track patients.

As there is no prior comparable registration of this, it is impossible to estimate a clinically relevant difference in order to make a power calculation and determine the amount of necessary registrations. Thus it has been decided that a 6-month registration will provide a reliable baseline. To avoid bias, the registration of this variable, will start after the end of the registration form period.

The overall aim of this study is, to ensure the best possible prehospital care for all stroke patients. The study will determine, if the EMD is at a high and international level in regards to stroke recognition, and if there is a potential to decrease on-scene time. This will serve as future comparison and have an effect on the structure and future education in the prehospital services, and potentially improve the outcome after acute ischemic stroke.

Distribution of responsibilities:

Søren Viereck; Medical student, University of Copenhagen; research employee/project manager: Literature search data analysis, development and evaluation of registration form for ambulance personnel, first draft of paper (planned 1. author) and fundraising.

Thea Palsgaard Møller; MD; Research fellow, Emergency Medical Services Copenhagen: Data extraction and supervision on data analysis, critical review of results.

Karl Bang Christensen: Associate Professor, Department of Biostatistics, University of Copenhagen: Critical review of protocol, supervision on statistical analyses, critical review of results.

Hanne Christensen; Senior Stroke Neurologist & Associate Professor, MD, PhD, DMSci, Department of Neurology, Bispebjerg Hospital, University of Copenhagen: Supervision, critical review of protocol, provision of data, supervision of data-analysis, critical review of results

Helle Klingenberg Iversen, MD, Senior Stroke Neurologist & associate professor Department of Neurology, Glostrup Hospital, University of Copenhagen: Supervision, critical review of protocol, provision of data, supervision of data-analysis, critical review of results.

Freddy Lippert; CEO, Emergency Medical Services in the Capital Region of Denmark; Associate professor, University of Copenhagen: Supervision, critical review of protocol, provision of data, supervision of data-analysis, critical review of results and overall clinical and scientific responsibility,

ELIGIBILITY:
Part 1.

Inclusion Criteria:

* All patients are included if registered in Danish Stroke Registry with an ICD-10 code of stroke (haemorrhagic and ischemic - I61 and I63-64.9), in the National Patient Registry with an ICD-10 code of TIA (Transient Ischemic Attack - G45.9) or in the Emergency Medical Services-database with a dispatch code of suspected stroke (A.26.03, A.26.04) from the 2-year period 01-01-2012 - 12-31-2013.

Exclusion Criteria:

* Patients are excluded if the Danish personal identification number is not available in either database. If the patient has been directly referred to the hospital by their general practitioner without the use of a EMS transport, or they have presented themselves in the emergency room, they will not be registered in the EMS database.

Part 2.

Inclusion Criteria:

* Patients with suspected stroke where the EMS has been in contact with fast track stroke service at the stroke centre are included.

Exclusion Criteria:

* Incomplete forms will be excluded.

Part 3.

Inclusion Criteria:

* All patients with a Danish personal identification number, referred to one of the two regional stroke centres, during a 6-month period will be included. The 6 month period will begin after the above mentioned 500 registration form has been collected, to avoid bias.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients suffering from a stroke in the Capital Region of Denmark. The Capital Region of Denmark is home to 1,8 mio. people and covers an area of 2.568 km². The regions has 24-hour fast track stroke service divided at 2 hospitals, with alternate 24-hour shifts.
Sampling Method: Probability Sample
Enrollment: 2653 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The rate of acute stroke recognized by the EMD during the emergency call (sensitivity). | 01.01.2012 - 12.31.2013 (up to 24 months)
Time from dispatch to ambulance arrival at the scene of accident in stroke fast track patients. | Up to 6 month period after collection of registration forms (expected 01.01.2015-06.30.2015)
Time on scene by EMS in stroke fast track patients (on-scene-time). | Up to 6 month period after collection of registration forms (expected 01.01.2015-06.30.2015)
Time from departure from the scene of the accident to arrival at the stroke centre in stroke fast track patients. | Up to 6 month period after collection of registration forms (expected 01.01.2015-06.30.2015)

SECONDARY OUTCOMES:
Final diagnoses(ICD-10), in patients with a dispatch code of stroke, but another final diagnosis (false positive). | 01.01.2012 - 12.31.2013 (up to 24 months)
Dispatch codes, in patients with a final diagnosis of acute stroke, but another dispatch code (false negative). | 01.01.2012 - 12.31.2013 (up to 24 months)
The positive predictive values of stroke recognition by healthcare personnel at the EMD. | 01.01.2012 - 12.31.2013 (up to 24 months)
The proportion of patients with a final diagnosis of stroke, who accessed the healthcare system through the EMS. | 01.01.2012 - 12.31.2013 (up to 24 months)
Prehospital time compared to in-hospital time in stroke fast track patients. | Up to 6 month period after collection of registration forms (expected 01.01.2015-06.30.2015)
Recognition of stroke by EMD in relation to treatment decisions in stroke fast track patients | Up to 6 month period after collection of registration forms (expected 01.01.2015-06.30.2015)

OTHER OUTCOMES:
On-scene-time in relation to time-point of performing 12-lead ECG | Up to 12 months.
  Will the time-point of performing 12-lead ECG (e.g. prior to departure) affect the on-scene-time?
On-scene-time in relation to quality of communication during prenotification of the stroke centre. | Up to 12 months.
  Will the quality of the communication during prenotification of the stroke centre, affect on-scene time?
On-scene-time in relation to ambulance operator | Up to 12 months.
  Will it affect on-scene-time, what company that operates the ambulance?
On-scene-time in relation to visitation to stroke fast track service | Up to 12 months.
  Will it affect the on-scene time, whether or not the patient is visitated to stroke fast track service?
On-scene-time in relation time-point of providing IV-accesses | Up to 12 months.
  Will the time-point of providing IV-accesses affect the on-scene time?
On-scene-time in relation to relatives being on the ambulance | Up to 12 months.
  Will it affect on-scene-time if relatives are accompanying the patient in the ambulance?
On-scene-time in relation to patients vomiting | Up to 12 months.
  Will it affect on-scene-time if a patient vomits?
Total on-scene-time in relation to specific time-intervals (se description) | Up to 12 months.
  This composite measure will determine if any of the following time-intervals are related to on-scene time.
  * Clinical tasks; including prior medical history, clinical examination and measurement of vital parameters
  * Communication in relation to prenotification of the stroke centre
  * Mobilization of the patient and on-scene conditions
  * Patient preparation; including IV-accesses and 12-lead ECG
On-scene-time in relation to ambulance manning | Up to 12 months.
  Will it affect on-scene-time, what manning that is on the ambulance?

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Lippert, MD, CEO, Study Director — Emergency Medical Services, Capital Region, Denmark
Locations (1):
- EMS Copenhagen, Copenhagen, Ballerup, Denmark

REFERENCES:
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group; Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 2010 May 15;375(9727):1695-703. doi: 10.1016/S0140-6736(10)60491-6. PMID 20472172
- [Background] Tong D, Reeves MJ, Hernandez AF, Zhao X, Olson DM, Fonarow GC, Schwamm LH, Smith EE. Times from symptom onset to hospital arrival in the Get with the Guidelines--Stroke Program 2002 to 2009: temporal trends and implications. Stroke. 2012 Jul;43(7):1912-7. doi: 10.1161/STROKEAHA.111.644963. Epub 2012 Apr 26. PMID 22539544
- [Background] Lin CB, Peterson ED, Smith EE, Saver JL, Liang L, Xian Y, Olson DM, Shah BR, Hernandez AF, Schwamm LH, Fonarow GC. Emergency medical service hospital prenotification is associated with improved evaluation and treatment of acute ischemic stroke. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):514-22. doi: 10.1161/CIRCOUTCOMES.112.965210. Epub 2012 Jul 10. PMID 22787065
- [Derived] Drenck N, Viereck S, Baekgaard JS, Christensen KB, Lippert F, Folke F. Pre-hospital management of acute stroke patients eligible for thrombolysis - an evaluation of ambulance on-scene time. Scand J Trauma Resusc Emerg Med. 2019 Jan 9;27(1):3. doi: 10.1186/s13049-018-0580-4. PMID 30626404
- [Derived] Viereck S, Moller TP, Iversen HK, Christensen H, Lippert F. Medical dispatchers recognise substantial amount of acute stroke during emergency calls. Scand J Trauma Resusc Emerg Med. 2016 Jul 7;24:89. doi: 10.1186/s13049-016-0277-5. PMID 27388490